CLINICAL TRIAL: NCT01802320
Title: A Phase 2 Study of MK-2206 in Previously Treated Metastatic Colorectal Cancer Patients Enriched for PTEN Loss and PIK3CA Mutation
Brief Title: Akt Inhibitor MK2206 in Treating Patients With Previously Treated Colon or Rectal Cancer That is Metastatic or Locally Advanced and Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-00487; NCI-2013-00487 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2012-0431 (Other: M D Anderson Cancer Center); 9340 (Other: CTEP); N01CM00039 (NIH); P30CA016672 (NIH)
Record Dates: First submitted 2013-02-27; First posted 2013-03-01 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-08

CONDITIONS: Colon Mucinous Adenocarcinoma; Colon Signet Ring Cell Adenocarcinoma; Rectal Mucinous Adenocarcinoma; Rectal Signet Ring Cell Adenocarcinoma; Recurrent Colon Carcinoma; Recurrent Rectal Carcinoma; Stage IIIA Colon Cancer; Stage IIIA Rectal Cancer; Stage IIIB Colon Cancer; Stage IIIB Rectal Cancer; Stage IIIC Colon Cancer; Stage IIIC Rectal Cancer; Stage IVA Colon Cancer; Stage IVA Rectal Cancer; Stage IVB Colon Cancer; Stage IVB Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — MK 2206

ARMS (1):
- Treatment (Akt inhibitor MK2206) (Experimental): Akt inhibitor MK2206 orally (PO) on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 24 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Akt Inhibitor MK2206; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: Akt Inhibitor MK2206 — Given PO
  Other Names: MK2206
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase II trial studies how well v-akt murine thymoma viral oncogene homolog 1 (Akt) inhibitor MK2206 works in treating patients with previously treated colon or rectal cancer that has spread from the primary site to other places in the body or nearby tissue or lymph nodes and cannot be removed by surgery. Akt inhibitor MK2206 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the response rate to MK-2206 (Akt inhibitor MK2206), defined as complete response (CR) + partial response (PR).

SECONDARY OBJECTIVES:

I. To determine response rate to MK-2206 in patients with phosphatase and tensin homolog (PTEN) loss or phosphatidylinositol-4,5-bisphosphate 3-kinase, catalytic subunit alpha (PIK3CA) mutation in a pretreatment biopsy from a metastatic site.

II. To determine progression-free survival (PFS) and overall survival (OS). III. To determine the time to treatment failure (TTF), and duration of tumor response (DR).

IV. To determine the safety profile and tolerability of this regimen in this patient population.

V. To determine effect of PTEN, v-raf murine sarcoma viral oncogene homolog B1 (BRAF), PIK3CA, and AKT mutations and semi-quantitative grading of PTEN expression on clinical response.

OUTLINE:

Patients receive Akt inhibitor MK2206 orally (PO) on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 24 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed, radiologically measurable metastatic or locally advanced unresectable colorectal adenocarcinoma that is amenable to image-guided biopsy; disease in previously radiated regions may not be considered measurable unless there has been demonstrated progression in the lesion
* Patients must have progressed on or been intolerant to a fluoropyrimidine-based chemotherapy regimen; there is no limit on the number of prior treatment regimens permitted
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Life expectancy of greater than 12 weeks
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< institution upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) =< 2.5 X institutional upper limit of normal or =< 5 X institutional upper limit of normal for patients with known liver metastasis
* Creatinine =< institution upper limit of normal OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Women of child-bearing potential and men must agree to use adequate contraception (double barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and 4 months after completion of MK-2206 administration; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of MK-2206 administration
* Patients must be able to swallow whole tablets; nasogastric or gastrostomy (G) tube administration is not allowed; tablets must not be crushed or chewed
* Ability to understand and the willingness to sign a written informed consent document
* Tumor must be wild type for the v-Ki-ras2 Kirsten rat sarcoma viral oncogene homolog (KRAS) and BRAF oncogenes, and must have known PIK3CA, AKT mutation status and PTEN expression status

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study; if the patient has residual toxicity from prior treatment, toxicity must be =< grade 1 (or =< grade 2 for peripheral neuropathy and/or alopecia)
* Patients who are receiving or have received any other investigational agents within 30 days of study day 1, or who have previously received MK-2206 at any time
* Patient has known active central nervous system (CNS) metastases and/or carcinomatous meningitis; however, patients with CNS metastases who have completed a course of therapy would be eligible for the study provided they are clinically stable for at least 1 month prior to entry as defined as:

  * No evidence of new or enlarging CNS metastasis
  * Off steroids that are used to minimize surrounding brain edema
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to MK-2206
* Patients receiving any medications or substances that are inhibitors or inducers of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP450 3A4) are ineligible
* Patients with diabetes or in risk for hyperglycemia should not be excluded from trials with MK-2206, but the hyperglycemia should be well controlled on oral agents before the patient enters the trial
* Cardiovascular baseline corrected QT by Fridericia's (QTcF) > 450 msec (male) or QTcF > 470 msec (female) will exclude patients from entry on study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with MK-2206
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for five years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edmund Kopetz, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: March 07, 2013 to July 14, 2015. All recruitment done at The University of Texas MD Anderson Cancer Center.
Groups:
- Treatment (Akt Inhibitor MK2206): Akt inhibitor MK2206 orally on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 24 months in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Treatment (Akt Inhibitor MK2206)
Started | 18
Completed | 16
Not Completed | 2
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 18
Age, Continuous [Median (Full Range); unit: years] | 56 [29 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 13
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (CR+PR) Evaluated Using Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: Complete Response (CR): Disappearance all target lesions. Any pathological lymph nodes must have reduction in short axis to <10 mm. Partial Response (PR): > 30% decrease in sum diameters of target lesions, reference baseline sum diameters. Progressive Disease (PD): > 20% increase in sum diameters of target lesions, reference smallest sum on study (includes baseline sum if smallest on study). In addition to relative increase of 20%, sum must demonstrate absolute increase of >5 mm. (Note: appearance of 1/> new lesions also considered progressions). Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, reference smallest sum diameters while on study.
Time Frame: Up to 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 18
Participants | 0

2. Secondary Outcome: Duration of Tumor Response (DR)
Description: Estimated using the Kaplan and Meier product limit method. Cox proportional hazards regression model will be used to identify prognostic factors for DR.
Time Frame: From the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented, assessed up to 18 months
Population: Outcome data not collected, no analysis to be performed as participants had related tumor response.
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Survival (OS)
Description: Estimated using the Kaplan and Meier product limit method. Cox proportional hazards regression model will be used to identify prognostic factors for OS.
Time Frame: Up to 18 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 18
months | 6.8 [5.83 to 7.77]

4. Secondary Outcome: Progression-free Survival (PFS)
Description: Estimated using the Kaplan and Meier product limit method. Cox proportional hazards regression model will be used to identify prognostic factors for PFS.
Time Frame: From start of treatment to time of progression or death, whichever occurs first, assessed up to 18 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 18
months | 1.87 [1.83 to 1.90]

5. Other Pre Specified Outcome: Validation of the Enrichment Biomarker Signature in Metastatic Sites
Description: Samples will be analyzed using the Wilcoxon rank test. Chi-square or Fisher's exact test where appropriate will be used to determine whether high levels of marker expression correlate with PTEN status.
Time Frame: Up to 18 months
Population: Given the lack of response seen in this study, biomarker validation and correlation of biomarker enrichment with clinical outcome is not feasible. Data were not collected.
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data collected during active 28 day cycle, treatment may continue for up to 24 months
Arm/Group | Treatment (Akt Inhibitor MK2206)
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 5/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Akt Inhibitor MK2206) (N=18)
Small Bowel Obstruction (Gastrointestinal disorders) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 1 (1)
Fracture, Arm (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Akt Inhibitor MK2206) (N=18)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Acute kidney injury (Injury, poisoning and procedural complications) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 1 (1)
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 7 (9)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anal pain (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 6 (10)
Anorexia (Metabolism and nutrition disorders) | 4 (6)
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 5 (7)
Blurred vision (Eye disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Creatinine increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 10 (12)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (4)
Dysarthria (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Eye disorders - (Other (Eye disorders) | 1 (2)
Fatigue (General disorders) | 7 (9)
Fever (General disorders) | 3 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Floaters (Eye disorders) | 1 (1)
Flu like symptoms (General disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Gait disturbance (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 11 (17)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (4)
Hypertension (Vascular disorders) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (3)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Lactate dehydrogenase (LDH) elevated (Investigations) | 1 (1)
Metabolism and nutrition disorders - (Other) (Metabolism and nutrition disorders) | 1 (1)
Mucosal infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Mucositis oral (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (1)
Nail ridging (Skin and subcutaneous tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 10 (14)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Progressive Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8)
Neutrophil count decreased (Investigations) | 1 (1)
Pain (General disorders) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Pharyngitis (Infections and infestations) | 1 (1)
Platelet count decreased (Investigations) | 4 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10 (11)
Blood Urea Nitrogen elevated (Renal and urinary disorders) | 1 (1)
Skin and subcutaneous tissue disorders - (Other) (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (3)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (6)
Weight loss (Investigations) | 4 (5)
Chloride decreased (Investigations) | 1 (2)
Platelet increased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less